CLINICAL TRIAL: NCT00418743
Title: A Phase II Randomised Trial of Second-line Treatment in Patients With Small Cell Lung Cancer (SCLC), Comparing Oral Combination Chemotherapy (CCNU, Cyclophosphamide, Etoposide) With Intravenous Association Chemotherapy.
Brief Title: Second-line Treatment in Patients With Small Cell Lung Cancer (SCLC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Collaborators: Baxter Healthcare Corporation (Industry); Amgen (Industry)
Responsible Party: Pr CHOUAID, GFPC
Other Study IDs: GFPC 05-01
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Small Cell Lung Cancer
Keywords: cancer; Lung cancer; small-cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine treatment efficacy and tolerability of second-line treatment in patients with small cell lung cancer comparing oral combinaison chemotherapy with intravenous combination chemotherapy.

DETAILED DESCRIPTION:
Determined treatment efficacy and tolerability of second-line treatment in patients with small cell lung cancer comparing oral combinaison chemotherapy with intravenous combination chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Small-cell lung cancer.
* Patients who, after (at least) a first line of chemotherapy based on platinum, had a partial response and then progressed, or who had a complete response and then relapsed within three months following the last course of this first-line therapy.
* Measurable or assessable disease.
* Life expectancy >2 months.
* Patients with a therapeutic risk level of <5 points (see section 6: "Treatment flowchart").
* Age >18 years;
* Performance status (WHO) <2;
* One measurable target lesion in a non irradiated region;
* Prior radiotherapy authorized unless it targeted the only measurable lesion;
* Biological criteria: WBC >2000/mm3, PMN >1500/mm3, platelets >100 000/mm3, creatinemia <2 x ULN, bilirubinemia <ULN, ALT and AST <2.5 x ULN (< 5 N if liver metastases)
* normal ECG
* written informed consent.

Exclusion Criteria:

* Non small-cell lung cancer.
* No objective response to platinum-based therapy
* Complete response lasting more than three months after the last course of first-line treatment.
* Symptomatic brain metastases.
* Bone metastases, carcinomatous lymphangitis, ascites or pleurisy as sole assessable disease manifestations.- Concurrent participation in another clinical trial.
* Therapeutic risk level of 6 points or more (see table)
* Uncontrolled clotting disorders;
* Uncontrolled severe infection;
* History of another malignancy, except for cervical carcinoma in situ or basocellular cancer that are considered cured;
* Psychological, familial, sociological or geographic circumstances preventing treatment follow-up as defined in the protocol;
* Patients deprived of their rights for administrative or legal reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Small-cell lung cancer who, after (at least) a first line of chemotherapy based on platinum, had a partial response and then progressed, or who had a complete response and then relapsed within three months following the last course of this first-line therapy.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2005-12; Study Completion 2010-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christos CHOUAID, Professor, Principal Investigator — Groupe Francais De Pneumo-Cancerologie
Locations (24):
- France (24):
  - Centre Hospitalier Universitaire, Angers
  - Site 05, Bastia
  - Site 22, Beauvais
  - Centre Hospitalier du Morvan, Brest
  - Centre François Baclesse, Caen
  - Site 43, Caen
  - Centre Hospitalier René Dubos, Cergy-Pontoise
  - Site 33, Créteil
  - Site 07, Draguignan
  - Site 32, Elbeuf
  - Site 04, Gap
  - Centre Hospitalier Les Oudairies, La Roche-sur-Yon
  - Hospital du Cluzeau, Limoges
  - Centre Hospitalier Régional, Longjumeau
  - Centre Hospitalier Lyon Sud, Lyon
  - Site 25, Mantes-la-Jolie
  - Site 06, Marseille
  - Site 27, Martigues
  - Site 01, Meaux
  - Hospital Saint Antoine, Paris
  - Site 17, Rouen
  - Hôpital Yves Le Foll, Saint-Brieuc
  - Site 14, Toulon
  - Site 11, Villefranche-sur-Saône

REFERENCES:
- See also: Groupement Francais de Pneumo-cancérologie — http://www.g-f-p-c.org